CLINICAL TRIAL: NCT01668199
Title: An Open-Label, Single-Dose, Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery and Pharmacokinetics of 14C TZP-101
Brief Title: A Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery and Pharmacokinetics of 14C TZP-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPJ5004-03/2011 (MET)
Record Dates: First submitted 2012-08-08; First posted 2012-08-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — ulimorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C TZP-101 (Experimental)
  Interventions: Drug: TZP-101

INTERVENTIONS:
Drug: TZP-101

SUMMARY:
A study to investigate the mass balance recovery and pharmacokinetics of 14C TZP-101.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males
* 35-65 years of age
* Body Mass Index (BMI) of 18-32 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Body weight of 75-90kg
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Subject must agree to use adequate methods of contraception

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 moths or more than 3 studies within the previous 12 months
* Participation in an ADE study within the previous 12 months
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption >21 units per week
* Current smokers and those who have smoked within the last 12 months, or a breath carbon monoxide (CO) reading of greater than 10ppm at screening
* Radiation exposure from clinical studies, including that from the present study, excluding background radiation including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Clinically significant abnormal biochemistry, haematology or urinalysis at screening as judged by the investigator
* Clinically significant abnormal physical findings, ECG or vital signs measurements at screening
* PR interval 220 ms at screening or on admission
* QTcB >450 ms at screening or on admission
* Existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the IMP
* History or presence of significant cardiovascular, respiratory, gastrointestinal (especially peptic ulcer disease), neurological, psychiatric, metabolic, hepatic or renal problems as judged by the investigator
* Positive drugs of abuse test result
* Positive HBV, HCV or HIV results
* Use of prescription or non prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 14 days of the planned IMP administration unless in the opinion of the PI the medication will not interfere with study procedures or compromise study safety
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of allergy requiring treatment (seasonal allergic rhinitis (hayfever) is allowed unless it is active)
* Donation or loss of greater than 400 mL of blood within the previous three months
* Subjects receiving or requiring prohibited medication as described in Section 11
* Failure to satisfy the Investigator of fitness to participate for any other reason
* Poor venous access

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of total radioactivity in plasma | 6 weeks
  To determine the pharmacokinetics of total radioactivity in plasma (Cmax, tmax, AUC, t1/2)
Pharmacokinetics of parent TZP-101 in plasma | 6 weeks
  To determine the pharmacokinetics of parent TZP-101 in plasma (Cmax, tmax, AUC, t1/2)
Total radioactivity in urine and faeces | 6 weeks
  To determine the Urine and faecal recovery of total radioactivity (Ae, Fe%, CLr)

SECONDARY OUTCOMES:
Total radioactivity in plasma | 6 weeks
  To determine the Total radioactivity in plasma/total radioactivity in whole blood ratio at selected timepoints
Total radioactivity of parent drug in plasma | 6 weeks
  To determine the Total radioactivity in plasma/parent drug in plasma ratio for selected PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MD, Principal Investigator — Quotient Clinical, Mere Way, Ruddlington Fields, Nottingham
Locations (1):
- Quotient Clinical, Nottingham, England, United Kingdom